CLINICAL TRIAL: NCT05277792
Title: Dosage of Tacrolimus Metabolites in Blood and Bile for Prediction of Its Side Effects in Liver Transplant Recipients
Acronym: STABILE 2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_8890_STABILE 2
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Blood Concentration of Tacrolimus Metabolites
Keywords: Tacrolimus, metabolites, liver transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate if concentration of tacrolimus metabolites is increased in patients presenting tacrolimus (TAC) side effects.

DETAILED DESCRIPTION:
The study will evaluate whether the blood concentration of TAC metabolites (13-O-desmethyl-tacrolimus, 15-O-desmethyl-tacrolimus and 31-O-desmethyl-tacrolimus), measured between Day1 and Day5 of its introduction, is increased in patients with TAC toxicity.

A blood test will be performed daily from Day1 to Day5 for the measurement of TAC concentration and TAC metabolites concentration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years) of both sexes,
* Candidates for liver transplantation or retransplantation, whatever the etiology and severity of the underlying disease,
* Not having expressed their opposition to participation in the study

Exclusion Criteria:

* Associated transplantation of another organ
* Contraindications to TAC administration
* Delayed introduction of TAC (beyond the 5th postoperative day) whatever the cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2022-05-08 (Actual); Primary Completion 2024-06-08 (Estimated); Study Completion 2024-06-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of blood concentration of TAC metabolites between patients presenting TAC related side effects or not. | Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No